CLINICAL TRIAL: NCT04012931
Title: A Phase 2, Open-label, Single-arm, Multicenter Study to Evaluate the Pharmacokinetics, Safety, Tolerability, and Efficacy of Switching to RPV Plus Other ARVs in HIV-1-infected Children (Aged 2 to <12 Years) Who Are Virologically Suppressed
Brief Title: A Study of Switching to RPV Plus Other ARVs in HIV-1-infected Children (Aged 2 to <12 Years) Who Are Virologically Suppressed
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108606; 2018-004301-32 (EudraCT Number); TMC278HTX2002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-07-08; First posted 2019-07-09 (Actual); Results first posted 2024-05-02 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: HIV
MeSH Terms: interventions — Rilpivirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Rilpivirine (RPV) (25 mg or adjusted weight-based dose) (Experimental): Participants will receive rilpivirine (RPV 25 milligram [mg], adjusted weight-based dose) orally once daily in combination with an investigator selected background regimen (that is investigator-selected antiretrovirals [ARVs] such as nucleoside/nucleotide reverse transcriptase inhibitor [N{t}RTIs] and integrase inhibitors) for 48 weeks.
  Interventions: Drug: Rilpivirine; Drug: ARV Background Regimen

INTERVENTIONS:
Drug: Rilpivirine — Rilpivirine 25 mg tablets for the 25 mg daily dose, or tablets for or a weight-adjusted dose. Administered orally once daily.
  Other Names: TMC278
Drug: ARV Background Regimen — The investigator-selected ARVs, including but not limited to N(t)RTIs (example, azidothymidine [AZT], abacavir [ABC], tenofovir alafenamide [TAF], or tenofovir disoproxil fumarate [TDF] in combination with emtricitabine [FTC] or lamivudine [3TC]), whichever are approved and marketed or considered local standard of care for children aged between 2 and < 12 years in a particular country are to be administered. Integrase inhibitors (for example, dolutegravir [DTG] or raltegravir) can also be administered in combination with RPV, as appropriate.

SUMMARY:
The purpose of this study is to evaluate the steady state pharmacokinetics (PK) of rilpivirine (RPV) and determine the appropriate dose of RPV in combination with other antiretrovirals (ARVs) in participants aged greater than or equal to 2 to less than 12 years and to evaluate the safety and tolerability of RPV in combination with other ARVs in participants of same age group over a 48-week treatment period with primary endpoint at Week 24.

DETAILED DESCRIPTION:
Participants infected with human immunodeficiency virus type 1 (HIV-1) are routinely treated with combinations of multiple drugs which reduces HIV-1 ribonucleic acid (RNA) to undetectable levels in a substantial proportion of participants and counteracts the risk of viral resistance development. RPV is a potent non-nucleoside reverse transcriptase inhibitor (NNRTI) with in vitro activity against wild type (WT) HIV-1 and against NNRTI-resistant HIV-1 mutants. A medical need still exists for the development of age/weight appropriate formulations in children less than (<) 12 years of age. In this study, participants will switch to RPV plus other ARVs. The primary analysis will be performed at Week 24. A participant will be considered to have completed the study if he or she has completed assessments at Week 48 of the study intervention phase. The total study duration for each participant, including screening and study intervention phases, will be approximately 54 weeks. Key efficacy assessments include determination of plasma HIV-1 RNA viral load and measurement of CD4+ cell count. Key safety assessments will include the monitoring of (serious) adverse events ([S]AEs) and HIV-related events, clinical laboratory tests, cardiovascular safety monitoring (vital signs and 12 lead electrocardiogram [ECGs]), and physical examination (including growth).

ELIGIBILITY:
Inclusion Criteria:

* Weighing at least 10 kilogram (kg) at screening
* Have documented chronic Human Immunodeficiency Virus (HIV-1) infection
* On a stable antiretroviral (ARV) regimen for at least 6 months prior to screening and virologically suppressed with documented evidence of at least 2 plasma viral loads less than (<) 50 HIV-1 ribonucleic acid (RNA) copies/milliliter (mL): one within 2-12 months prior to screening and one at screening
* Can switch from any ARV class
* Never been treated with a therapeutic HIV vaccine
* Historical HIV-1 genotyping result at screening for children aged >=2 to <6 years (and for children aged >=6 to <12 years if a historical HIV-1 genotyping result is available at screening) must demonstrate sensitivity to RPV and to the selected background ARVs

Exclusion Criteria:

* Have previously documented HIV-2 infection
* Have known or suspected acute (primary) HIV-1 infection
* Taken any disallowed concomitant therapies within 4 weeks before the planned first dose of study intervention
* Any current or history of adrenal disorder
* A history of virologic failure to ARVs with or without availability of an HIV-1 genotype result at the time of failure

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (14):
- Italy (3):
  - ASST Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - IRCCS Ospedale Pediatrico Bambino Gesu, Roma
- Portugal (2):
  - Uls Santa Maria - Hosp. Santa Maria, Lisbon
  - Uls Sao Joao - Hosp. Sao Joao, Porto
- South Africa (2):
  - Josha Research, Bloemfontein
  - Family Clinical Research Unit FAM-CRU, Tygerberg
- Spain (3):
  - Hosp. Sant Joan de Deu, Esplugues de Llobregat
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. La Paz, Madrid
- Thailand (3):
  - Siriraj Hospital Mahidol University, Bangkok
  - Research Institute for Health Sciences, Chiang Mai
  - Bamrasnaradura Infectious Disease Institute, Nonthaburi
- Joint Clinical Research Centre, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participant flow is based on the initial administered dose, irrespective of subsequent dose-alterations. Out of the 2 participants weighing <20 kg who received rilpivirine 15 mg, 1 participant switched to rilpivirine 12.5 mg group after the first 4 weeks. This participant was counted in the <20 kg rilpivirine 15 mg group in the Participant flow section, whereas it was counted in the <20 kg rilpivirine 12.5 mg group for the pharmacokinetic assessments reported in the outcome measure section.
Groups:
- Rilpivirine: Participants weighing less than (<) 20 kilograms (kg) received rilpivirine 12.5 milligrams (mg) or 15 mg; 20 to <25 kg received rilpivirine 15 mg; greater than equal to (>=) 25 kg received rilpivirine 25 mg orally once daily in combination with investigator-selected antiretrovirals (ARVs), including but not limited to nucleoside/nucleotide reverse transcriptase inhibitor (N[t]RTIs) (example, azidothymidine [AZT], abacavir [ABC], tenofovir alafenamide [TAF], or tenofovir disoproxil fumarate [TDF] in combination with emtricitabine [FTC] or lamivudine [3TC]), whichever were approved and marketed or considered local standard of care for children aged between >=2 and <12 years in a particular country. Integrase inhibitors (for example, dolutegravir [DTG] or raltegravir) were administered in combination with rilpivirine as appropriate. The overall treatment duration of the study was 52 weeks.
Period: Overall Study
Arm/Group | Rilpivirine
Started | 26
Participants Aged 2 to <6 Years | 1
Participants Aged >=6 to <12 Years | 25
Participants >=25 kg Who Received 25 mg Rilpivirine | 18
Participants 20 to <25 kg Who Received 15 mg Rilpivirine | 5
Participants <20 kg Who Received 15 mg Rilpivirine | 2
Participants <20 kg Who Received 12.5 mg Rilpivirine | 1
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Rilpivirine
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.5 (1.83)
Age, Customized [Count of Participants; unit: Participants]
  Children (2-12 years) | 26
  Adolescents (12-17 years) | 0
  Adults (18-64 years) | 0
  From 65 to 84 years | 0
  85 years and over | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Italy | 5
  Portugal | 1
  South Africa | 8
  Spain | 3
  Thailand | 7
  Uganda | 2

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time of Administration up to 24 Hours Postdose (AUC[0-24h]) of Rilpivirine 12.5 mg (for <20 kg Group)
Description: AUC(0-24h) was defined the area under the plasma concentration-time curve from time of administration up to 24 hours postdose of rilpivirine. As planned, data was not summarized for arms where number of participants analyzed was less than 3. Only individual participant data was available and reported in this outcome measure. Out of the 2 participants weighing <20 kg who received rilpivirine 15 mg, 1 participant switched to rilpivirine 12.5 mg group after the first 4 weeks. This participant was counted in the <20 kg rilpivirine 12.5 mg group for the pharmacokinetic assessments, hence the number of participants analyzed for this outcome measure in this arm are exceeding the participants that started this arm. As per protocol, the intensive PK samples were collected at anytime during Day 28 to Day 32 after first dose at the specified dose regimen.
Time Frame: Predose up to 24 hour post-dose at anytime during Day 28 to Day 32 (Week 4)
Population: Full analysis set (FAS): who had taken at least 1 dose of rilpivirine. N (number of participants analyzed): who were evaluable for this outcome measure, intensive PK data was collected from a subset of participants.
Measure: Mean (Standard Deviation); unit: nanograms*hour/milliliter (ng*h/mL)
Groups:
- Rilpivirine 12.5 Milligrams (mg) (<20 kg): Participants weighing less than (<)20 kilograms (kg) received rilpivirine 12.5 mg orally once daily in combination with investigator-selected background regimen, that were approved and marketed or considered local standard of care for children aged between 2 and 12 years in a particular country.
Arm/Group | Rilpivirine 12.5 Milligrams (mg) (<20 kg)
Number analyzed (Participants) | 2
nanograms*hour/milliliter (ng*h/mL)
  Participant 1: number analyzed (Participants) | 1
  Participant 1 | 4116 (NA) — Standard deviation could not be calculated for a single participant.
  Participant 2: number analyzed (Participants) | 1
  Participant 2 | 4646 (NA) — Standard deviation could not be calculated for a single participant.

2. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time of Administration up to 24 Hours Postdose (AUC[0-24h]) of Rilpivirine 15 mg (for <20 kg Group)
Description: AUC(0-24h) was defined the area under the plasma concentration-time curve from time of administration up to 24 hours postdose of rilpivirine. As per protocol, the intensive PK samples were collected at anytime during Day 28 to Day 32 after first dose at the specified dose regimen.
Time Frame: Predose up to 24 hour post-dose at anytime during Day 28 to Day 32 (Week 4)
Population: FAS included all participants who had taken at least 1 dose of rilpivirine. N (number of participants analyzed): who were evaluable for this outcome measure, intensive PK data was collected from a subset of participants.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Groups:
- Rilpivirine 15 mg (<20 kg): Participants weighing <20 kg received rilpivirine 15 mg orally once daily in combination with investigator-selected background regimen, whichever were approved and marketed or considered local standard of care for children aged between 2 and 12 years in a particular country.
Arm/Group | Rilpivirine 15 mg (<20 kg)
Number analyzed (Participants) | 1
ng*h/mL | 3494 (NA) — Standard deviation could not be calculated for a single participant.

3. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time of Administration up to 24 Hours Postdose (AUC[0-24h]) of Rilpivirine 15 mg (for 20 to <25 mg Group)
Description: as for outcome 2
Time Frame: Predose up to 24 hour post-dose at anytime during Day 28 to Day 32 (Week 4)
Population: FAS included all participants who had taken at least 1 dose of rilpivirine.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Groups:
- Rilpivirine 15 mg (20 to <25 kg): Participants weighing 20 to <25 kg received rilpivirine 15 mg orally once daily in combination with investigator-selected background regimen, whichever were approved and marketed or considered local standard of care for children aged between 2 and 12 years in a particular country.
Arm/Group | Rilpivirine 15 mg (20 to <25 kg)
Number analyzed (Participants) | 5
ng*h/mL | 3506 (946)

4. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time of Administration up to 24 Hours Postdose (AUC[0-24h]) of Rilpivirine 25 mg (for >=25 kg Group)
Description: AUC(0-24h) was defined the area under the plasma concentration-time curve from time of administration up to 24 hours postdose of rilpivirine. As planned, data was not summarized for arms where number of participants analyzed was less than 3. Only individual participant data was available and reported in this outcome measure. As per protocol, the intensive PK samples were collected at anytime during Day 28 to Day 32 after first dose at the specified dose regimen.
Time Frame: Predose up to 24 hour post-dose at anytime during Day 28 to Day 32 (Week 4)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*h/mL
Groups:
- Rilpivirine 25 mg (>=25 kg): Participants weighing >=25 kg received rilpivirine 25 mg orally once daily in combination with investigator-selected background regimen, whichever were approved and marketed or considered local standard of care for children aged between 2 and 12 years in a particular country.
Arm/Group | Rilpivirine 25 mg (>=25 kg)
Number analyzed (Participants) | 2
ng*h/mL
  Participant 1: number analyzed (Participants) | 1
  Participant 1 | 4514 (NA) — Standard deviation could not be calculated for a single participant.
  Participant 2: number analyzed (Participants) | 1
  Participant 2 | 5644 (NA) — Standard deviation could not be calculated for a single participant.

5. Secondary Outcome: Percentage of Participants With HIV-1 Ribonucleic Acid (RNA) <50 and >=50 Copies/mL Through Weeks 24 and 48
Description: Percentage of participants with a HIV-1 RNA less than (<) 50 copies per mL and greater than or equal to (>=)50 copies/mL were assessed using Food and Drug Administration (FDA) snapshot approach which defines a participant's virologic response status using only the viral load at the predefined time point within a window of time, along with study drug discontinuation status. HIV-1 RNA level <50 copies per mL, was considered as virologic success and >= 50 copies/mL was considered as virological failure as per the snapshot approach. The FDA snapshot analysis at Week 24 and Week 48 was based on the last observed plasma viral load data within the visit window (that is, Weeks 24 and 48).
Time Frame: From Day 1 up to Weeks 24 and 48
Population: FAS included all participants who had taken at least 1 dose of rilpivirine.
Measure: Number; unit: Percentage of participants
Groups:
- Rilpivirine: >=2 to <6 Years: Participants weighing <20 kilograms (kg) received rilpivirine 12.5 milligrams (mg) or 15 mg; 20-<25 kg received 15 mg; >=25 kg received 25 mg orally once daily in combination with investigator-selected background regimen, whichever were approved and marketed or considered local standard of care for children aged between >=2 and <6 years in a particular country. Integrase inhibitors (for example, dolutegravir [DTG] or raltegravir) could also be administered in combination with rilpivirine as appropriate.
- Rilpivirine: >=6 to <12 Years: Participants weighing <20 kg received rilpivirine 12.5 mg or 15 mg; 20-<25 kg received 15 mg; >=25 kg received 25 mg orally once daily in combination with investigator-selected background regimen, whichever were approved and marketed or considered local standard of care for children aged between >=6 and <12 years in a particular country. Integrase inhibitors (for example, dolutegravir [DTG] or raltegravir) could also be administered in combination with rilpivirine as appropriate.
Arm/Group | Rilpivirine: >=2 to <6 Years | Rilpivirine: >=6 to <12 Years
Number analyzed (Participants) | 1 | 25
Percentage of participants
  Week 24: <50 copies/mL | 100.0 | 100.0
  Week 24: >=50 copies/mL | 0.0 | 0.0
  Week 48: <50 copies/mL | 100.0 | 100.0
  Week 48: >=50 copies/mL | 0.0 | 0.0

6. Secondary Outcome: Percentage of Participants With HIV-1 Ribonucleic Acid (RNA) <400 and >=400 Copies/mL Through Weeks 24 and 48
Description: Percentage of participants with viral load (plasma HIV-1 RNA levels) <400 copies/mL and >=400 copies/mL were assessed by the FDA snapshot approach which defines a participant's virologic response status using only the viral load at the predefined time point within a window of time, along with study drug discontinuation status. HIV-1 RNA level <400 copies per mL, was considered as virologic success and >=400 copies/mL was considered as virological failure as per the snapshot approach. The FDA snapshot analysis at Week 24 and Week 48 was based on the last observed plasma viral load data within the visit window (that is, Weeks 24 and 48).
Time Frame: From Day 1 up to Weeks 24 and 48
Population: FAS included all participants who had taken at least 1 dose of rilpivirine.
Measure: Number; unit: Percentage of participants
Arm/Group | Rilpivirine: >=2 to <6 Years | Rilpivirine: >=6 to <12 Years
Number analyzed (Participants) | 1 | 25
Percentage of participants
  Week 24: <400 copies/mL | 100.0 | 100.0
  Week 24: >=400 copies/mL | 0.0 | 0.0
  Week 48: <400 copies/mL | 100.0 | 100.0
  Week 48: >=400 copies/mL | 0.0 | 0.0

7. Secondary Outcome: Change From Baseline in Cluster of Differentiation 4 (CD4+) Cell Count up to Week 24 and Week 48
Description: The immunologic change was determined by changes in CD4+ cell count using non-completer = failure imputation, that was, missing values after discontinuation were imputed with the baseline value, thus resulting in a 0 change. For intermittent missing data, last observation carried forward (LOCF) approach was applied.
Time Frame: From baseline (Day 1) up to Weeks 24 and 48
Population: FAS included all participants who had taken at least 1 dose of rilpivirine.
Measure: Mean (Standard Error); unit: Cells/cubic millimeter
Arm/Group | Rilpivirine: >=2 to <6 Years | Rilpivirine: >=6 to <12 Years
Number analyzed (Participants) | 1 | 25
Cells/cubic millimeter
  Week 24 | 313.0 (NA) — Standard error could not be calculated for a single participant. | 26.3 (32.10)
  Week 48 | 279.0 (NA) — Standard error could not be calculated for a single participant. | -19.9 (28.52)

8. Secondary Outcome: Predose Plasma Concentration (C[0h]) of Rilpivirine 12.5 mg (for <20 kg Group)
Description: C(0h) was defined as the predose plasma concentration of rilpivirine. As planned, data was not summarized for arms where number of participants analyzed was less than 3. Only individual participant data was available and reported in this outcome measure. Out of the 2 participants weighing <20 kg who received rilpivirine 15 mg, 1 participant switched to rilpivirine 12.5 mg group after the first 4 weeks. This participant was counted in the <20 kg rilpivirine 12.5 mg group for the pharmacokinetic assessments, hence the number of participants analyzed for this outcome measure in this arm are exceeding the participants that started this arm. As per protocol, the intensive PK samples were collected at anytime during Day 28 to Day 32 after first dose at the specified dose regimen.
Time Frame: Predose at anytime during Day 28 to Day 32 (Week 4)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Rilpivirine 12.5 Milligrams (mg) (<20 kg)
Number analyzed (Participants) | 2
ng/mL
  Participant 1: number analyzed (Participants) | 1
  Participant 1 | 116 (NA) — Standard deviation could not be calculated for a single participant.
  Participant 2: number analyzed (Participants) | 1
  Participant 2 | 161 (NA) — Standard deviation could not be calculated for a single participant.

9. Secondary Outcome: Predose Plasma Concentration (C[0h]) of Rilpivirine 15 mg (for <20 kg Group)
Description: C(0h) was defined as the predose plasma concentration of rilpivirine. As per protocol, the intensive PK samples were collected at anytime during Day 28 to Day 32 after first dose at the specified dose regimen.
Time Frame: Predose at anytime during Day 28 to Day 32 (Week 4)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Rilpivirine 15 mg (<20 kg)
Number analyzed (Participants) | 1
ng/mL | 79.3 (NA) — Standard deviation could not be calculated for a single participant.

10. Secondary Outcome: Predose Plasma Concentration (C[0h]) of Rilpivirine 15 mg (for 20 to <25 kg Group)
Description: as for outcome 9
Time Frame: Predose at anytime during Day 28 to Day 32 (Week 4)
Population: FAS included all participants who had taken at least 1 dose of rilpivirine.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Rilpivirine 15 mg (20 to <25 kg)
Number analyzed (Participants) | 5
ng/mL | 138 (58.7)

11. Secondary Outcome: Predose Plasma Concentration (C[0h]) of Rilpivirine 25 mg (for >=25 kg Group)
Description: C(0h) was defined as the predose plasma concentration of rilpivirine. As planned, data was not summarized for arms where number of participants analyzed was less than 3. Only individual participant data was available and reported in this outcome measure. As per protocol, the intensive PK samples were collected at anytime during Day 28 to Day 32 after first dose at the specified dose regimen.
Time Frame: Predose at anytime during Day 28 to Day 32 (Week 4)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Rilpivirine 25 mg (>=25 kg)
Number analyzed (Participants) | 2
ng/mL
  Participant 1: number analyzed (Participants) | 1
  Participant 1 | 146 (NA) — Standard deviation could not be calculated for a single participant.
  Participant 2: number analyzed (Participants) | 1
  Participant 2 | 342 (NA) — Standard deviation could not be calculated for a single participant.

12. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Rilpivirine 12.5 mg (for <20 kg Group)
Description: Cmax was defined as the maximum observed plasma concentration of rilpivirine. As planned, data was not summarized for arms where number of participants analyzed was less than 3. Only individual participant data was available and reported in this outcome measure. Out of the 2 participants weighing <20 kg who received rilpivirine 15 mg, 1 participant switched to rilpivirine 12.5 mg group after the first 4 weeks. This participant was counted in the <20 kg rilpivirine 12.5 mg group for the pharmacokinetic assessments, hence the number of participants analyzed for this outcome measure in this arm are exceeding the participants that started this arm. As per protocol, the intensive PK samples were collected at anytime during Day 28 to Day 32 after first dose at the specified dose regimen.
Time Frame: Predose up to 24 hour post-dose at anytime during Day 28 to Day 32 (Week 4)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Rilpivirine 12.5 Milligrams (mg) (<20 kg)
Number analyzed (Participants) | 2
ng/mL
  Participant 1: number analyzed (Participants) | 1
  Participant 1 | 273 (NA) — Standard deviation could not be calculated for a single participant.
  Participant 2: number analyzed (Participants) | 1
  Participant 2 | 318 (NA) — Standard deviation could not be calculated for a single participant.

13. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Rilpivirine 15 mg (for <20 kg Group)
Description: Cmax was defined as the maximum observed plasma concentration of rilpivirine. As per protocol, the intensive PK samples were collected at anytime during Day 28 to Day 32 after first dose at the specified dose regimen.
Time Frame: Predose up to 24 hour post-dose at anytime during Day 28 to Day 32 (Week 4)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Rilpivirine 15 mg (<20 kg)
Number analyzed (Participants) | 1
ng/mL | 214 (NA) — Standard deviation could not be calculated for a single participant.

14. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Rilpivirine 15 mg (for 20 to <25 mg Group)
Description: as for outcome 13
Time Frame: Predose up to 24 hour post-dose at anytime during Day 28 to Day 32 (Week 4)
Population: FAS included all participants who had taken at least 1 dose of rilpivirine.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Rilpivirine 15 mg (20 to <25 kg)
Number analyzed (Participants) | 5
ng/mL | 217 (43.1)

15. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Rilpivirine 25 mg (for >=25 kg Group)
Description: Cmax was defined as the maximum observed plasma concentration of rilpivirine. As planned, data was not summarized for arms where number of participants analyzed was less than 3. Only individual participant data was available and reported in this outcome measure. As per protocol, the intensive PK samples were collected at anytime during Day 28 to Day 32 after first dose at the specified dose regimen.
Time Frame: Predose up to 24 hour post-dose at anytime during Day 28 to Day 32 (Week 4)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Rilpivirine 25 mg (>=25 kg)
Number analyzed (Participants) | 2
ng/mL
  Participant 1: number analyzed (Participants) | 1
  Participant 1 | 309 (NA) — Standard deviation could not be calculated for a single participant.
  Participant 2: number analyzed (Participants) | 1
  Participant 2 | 418 (NA) — Standard deviation could not be calculated for a single participant.

16. Secondary Outcome: Percentage of Participants With Viral Genotype at the Time of Virologic Failure at Weeks 24 and 48
Description: Percentage of participants with viral genotype at the time of virologic failure (that is, HIV 1 RNA >=50 copies/mL and >=400 copies/mL) per FDA snapshot approach were reported. Confirmed virologic failure was defined as 2 consecutive HIV-1 RNA plasma viral load measurements >=200 copies/mL and suspected virologic failure was defined as HIV-1 RNA >=200 copies/mL. No participant achieved virologic failure hence this outcome measure could not be evaluated.
Time Frame: Weeks 24 and 48
Population: FAS included all participants who had taken at least 1 dose of rilpivirine.
Arm/Group | Rilpivirine: >=2 to <6 Years | Rilpivirine: >=6 to <12 Years
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Percentage of Participants With Treatment Adherence >95% Based on Tablet Count up to Weeks 24 and 48
Description: Percentage of participants with treatment adherence greater than (>) 95 percent (%) as assessed by tablet count (study intervention accountability) up to Weeks 24 and 48 of study treatment were reported. Treatment adherence was defined as having a treatment adherence of >95% by tablet count.
Time Frame: From Day 1 up to Weeks 24 and 48
Population: FAS included all participants who had taken at least 1 dose of rilpivirine. N (number of participants analyzed): participants who were evaluable for this outcome measure. For participants who never returned kits dispensed at baseline, adherence could not be derived.
Measure: Number; unit: Percentage of participants
Arm/Group | Rilpivirine: >=2 to <6 Years | Rilpivirine: >=6 to <12 Years
Number analyzed (Participants) | 1 | 22
Percentage of participants
  Week 24 | 100.0 | 86.4
  Week 48 | 100.0 | 90.9

18. Secondary Outcome: Change From Baseline in Percentage of Cluster of Differentiation 4 (CD4+) Cell Count up to Week 24 and Week 48
Description: as for outcome 7
Time Frame: From baseline (Day 1) up to Weeks 24 and 48
Population: FAS included all participants who had taken at least 1 dose of rilpivirine.
Measure: Mean (Standard Error); unit: Percentage of lymphocytes
Arm/Group | Rilpivirine: >=2 to <6 Years | Rilpivirine: >=6 to <12 Years
Number analyzed (Participants) | 1 | 25
Percentage of lymphocytes
  Week 24 | 5.3 (NA) — Standard error could not be calculated for a single participant | 1.2 (1.04)
  Week 48 | 6.4 (NA) — Standard error could not be calculated for a single participant | 0.7 (1.14)

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) up to Week 52
Description: Safety was based on the full analysis set (FAS) which included all participants who had taken at least 1 dose of rilpivirine.
Arm/Group | Rilpivirine
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 11/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rilpivirine (N=26)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (3)
Vomiting (Gastrointestinal disorders) | 4 (16)
Pyrexia (General disorders) | 2 (2)
Rhinitis (Infections and infestations) | 2 (3)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2)
Alanine Aminotransferase Increased (Investigations) | 3 (5)
Aspartate Aminotransferase Increased (Investigations) | 2 (2)
Decreased Appetite (Metabolism and nutrition disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2021-02-22): https://cdn.clinicaltrials.gov/large-docs/31/NCT04012931/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-27): https://cdn.clinicaltrials.gov/large-docs/31/NCT04012931/SAP_001.pdf